CLINICAL TRIAL: NCT00001069
Title: A Randomized Study of the Clinical Effects of Initiating or Changing Antiretroviral Therapy Based on Plasma HIV RNA Quantitation Compared With Initiating or Changing Therapy Based on Current Clinical Practice Alone
Brief Title: A Study of Two Methods of Determining When to Begin or Change Anti-HIV Treatment
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: CPCRA 036
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-01

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Decision Making; Physician's Practice Patterns
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
PRIMARY: To compare the clinical efficacy of two decision making strategies for initiating or changing antiretroviral therapy: decision making based on current clinical practice alone (i.e., initiating or changing therapy based on CD4 count decline and/or clinical progression) versus decision making based on plasma HIV RNA quantitation in addition to current clinical practice.

SECONDARY: To evaluate toxicity, biological markers, and patient management in the two arms.

Although changing therapies is a common strategy in the treatment of HIV disease, guidelines are needed to help clinicians and patients decide when a change in antiretroviral therapy is indicated. The technology of measuring HIV RNA in plasma has been suggested as a tool for monitoring clinical drug efficacy. However, uncertainty remains about whether aggressive antiretroviral treatment to lower HIV RNA and maintain low levels for as long as possible will confer clinical benefit in comparison with management based on monitoring CD4 counts and HIV-related symptoms.

DETAILED DESCRIPTION:
Although changing therapies is a common strategy in the treatment of HIV disease, guidelines are needed to help clinicians and patients decide when a change in antiretroviral therapy is indicated. The technology of measuring HIV RNA in plasma has been suggested as a tool for monitoring clinical drug efficacy. However, uncertainty remains about whether aggressive antiretroviral treatment to lower HIV RNA and maintain low levels for as long as possible will confer clinical benefit in comparison with management based on monitoring CD4 counts and HIV-related symptoms.

Patients are randomized to a decision making strategy for initiating or changing therapy based on current clinical practice alone vs. decision making based on plasma HIV RNA quantitation in addition to current clinical practice in patients with <= 300 CD4+ cells/mm3. All patients in the RNA arm as well as a subset (n = 183) of those in the CCP arm will have a plasma HIV RNA quantitation drawn every 4 months. The results of these quantitations will be blinded until the end of the study. CD4 counts will be obtained at least every 4 months if the previous count was > 20 cells/mm3. The remaining patients in the CCP arm will have CD4 counts obtained according to their clinicians' current clinical practices. Medications, clinical status, and changes in antiretroviral therapy will be recorded for all patients in the study. Patients are stratified by CD4+ cell count (<100 cells/mm3 [200 patients] vs. 100-300 cells/mm3 [900 patients]).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 count <= 300 cells/mm3.
* NO stage 2 or worse AIDS dementia complex.
* Life expectancy of at least 6 months.
* Reasonably good health.
* age >= 13yrs.
* signed informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Disorders or conditions that may prevent adequate compliance with study requirements.

Patients with the following prior conditions are excluded:

* Stage 2 >= AIDS dementia complex.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100

CONTACTS AND LOCATIONS:
Overall Officials: Thompson M, Study Chair; Perez G, Study Chair
Locations (17):
- United States (17):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Baltimore Trials, Baltimore, Maryland
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners Research, Albuquerque, New Mexico
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Doepel LK. Volunteers needed for study of HIV viral load test. NIAID AIDS Agenda. 1995 Dec:3. PMID 11363351
- [Background] James JS. Viral load: new "strategy" trial in 15 U.S. cities. AIDS Treat News. 1995 Oct 20;(no 233):1-3. PMID 11363037
- [Background] Raghavan S, Grant LB, Barisch G, Thompson M, Williams B, Matoe N, el-Sadr WM. Change in log10 HIV RNA and protease inhibitor use associated with weight change in HIV+ men in a national clinical trial. Int Conf AIDS. 1998;12:556 (abstract no 32180)